CLINICAL TRIAL: NCT05075343
Title: The Effects of Custom-made Foot Orthoses on Foot Pain, Foot Function, Gait Function and Freeliving Walking Activities in Psoriatic Arthritis (PsA) Patients: A Pre-experimental Trial
Brief Title: Effect of Custom Foot Orthoses in Patients With Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Boissy (Other)
Responsible Party: Sponsor-Investigator, Patrick Boissy, Professor, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-3182
Record Dates: First submitted 2021-09-20; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Psoriatic Arthritis; Foot Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Custom foot orthoses (CFO) (Experimental): Participants with a confirmed diagnosis of PsA and foot pain received and wore custom foot orthoses (CFO).
  Interventions: Device: Custom foot orthoses

INTERVENTIONS:
Device: Custom foot orthoses — 3D printed custom foot orthoses (CFO) were designed by the same experimented podiatrist based on a detailed clinical and biomechanical examination and a 3D foot scan obtained for each participant. The degrees and types were adjusted at the CFO delivery according to each patient's comfort and tolerance.
  The intervention period was 7weeks. The participants were taught to wear the CFO progressively during the first two weeks to allow for the lower limbs' muscles and structures to adjust to the CFO, and to wear the orthoses for the next 5 weeks, 7 days a week as often as they could.

SUMMARY:
Foot involvement is a major concern in psoriatic arthritis (PsA). The patients could experience severe levels of foot pain and disability and reduced mobility and quality of life. Previous studies showed that the use of Custom foot orthoses (CFO) was effective to improve foot pain and perceived disability in patients with foot disease associated with rheumatoid arthritis. However, there are no records in the literature on the effectiveness of CFO in PsA patients. Therefore, our objective was o explore the effects of CFO on foot pain, foot function, gait spatiotemporal parameters (STP), and ambulatory physical activity (APA) in PsA patients with foot involvement.

In this pre-experimental exploratory study, 22 PsA patients having stable medication in the last 3 months preceding the recruitment were recruited. All the patients wore functional CFO designed by an experimented podiatrist during a 7-week period. Foot and lower limb pain and foot function were measured at baseline (T0) and after the 7-week period using the numerical rating scale (NRS) and the foot function index (FFI), respectively. Gait function was assessed by recording spatiotemporal parameters (STPs) during a 10-meter walk test using an instrumented gait analysis system (Mobility Lab) at T0 and T7. Freeliving walking activities (step count, freeliving cadence, time spent in different ambulatory physical activity (APA) intensities) at T0 and T7 were recorded over 7 days using accelerometer data collected from an instrumented sock worn by the participants during waking hours.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 70 years
* Diagnosed with psoriatic arthritis by a rheumatologist
* Having moderate to severe foot pain scored at least 3 on the numeric rating scale
* Having stable medication for the three months preceding the study

Exclusion Criteria:

* Having diabetes or neurological disease that may affect the feet
* Having recent traumatic foot injury
* Having received specific interventions for the feet (ex: foot orthoses, orthopedic shoes, intraarticular steroid injection) for the three months preceding the study.
* Having a recent history of foot surgery.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Foot function | up to 12 weeks
  Foot function was measure using the Foot function index (FFI). The FFI is a self-reported questionnaire composed of 23 items divided into three subscales measuring foot pain (FFI-P), foot disability (FFI-D) and foot-related activity limitation (FFI-AL). Each item of The FFI was recorded on a NRS (0 to 10) allowing for the calculation of both, total and subscale scores. The values range between 0 and 100, with higher values indicating greater pain, disability, and activity limitation.

SECONDARY OUTCOMES:
Foot pain | up to 12 weeks
  The intensity of foot pain was measured using a zero-to-ten numeric rating scale (NRS). Participants were asked to circle a number between 0 and 10 that fits best their average pain intensity at the foot in the seven days preceding data collection. Foot pain was assessed more in details (e.g. pain at walking with foot orthoses, pain at walking with shoes, pain at the end of the day etc.) with the pain sub-scale of the foot function index (FFI). Moreover, to monitor the evolution of weekly foot pain intensity during the intervention period, the patients were asked to record at the end of each week, the intensity of foot pain in a diary using 0 to 10 NRS.
Orthoses wearing time | 7 weeks
  Orthoses wearing time was assessed by asking the participants to record in a diary that included a calendar covering the 7-week intervention period, the daily wearing time in hours. The CFO wearing time is reported as the average wearing time per week.
Global and lower limb pain | up to 12 weeks
  Global pain and pain at the knee, hip, and lower back pain, were measured using the NRS (0, no pain - 10, worst imaginable pain).
Gait function | up to 12 weeks
  Gait function was assessed using an instrumented gait analysis system. Gait spatiotemporal parameters (STPs) including cadence, gait cycle duration, gait speed, stride length, double support, swing time, foot strike angle, and stride time variability, were recorded using the Mobility Lab system (APDM Wearable Technologies) during 10 meters walk test (10MWT). Mobility Lab is research grade system that has been proven to be accurate and reliable in estimating STP. Mobility Lab uses a set of six OPAL inertial measurement units (IMUs) and a software that allows for an automated and easy extraction of STP. All the participants performed three 10MWT trials over a 14-meters straight walkway with the Mobility lab's IMUs fixed with elastics straps on the chest, the lower back and both wrists and feet. The walks were performed at the participants' comfortable speed and the average of the three trials was calculated.
Freeliving walking activities | up to 12 weeks
  Freeliving walking activities including step count, freeliving cadence, and time spent in ambulatory physical activity (APA) intensity-based categories were assessed using an instrumented sock (Sensoria Inc, Redmond, WA, USA) with an embedded 9 axis IMU positioned at the ankle. The instrumented sock connects automatically, without any manipulation needed from the participants, via Bluetooth to a smartwatch (Apple Watch, series 3) where the raw inertial measures of motion (3D accelerometer) are stored and then transferred to a PC for data reduction and processing to extract gait activities specific outcomes.

OTHER OUTCOMES:
Control variables | 7 weeks
  The participants were asked to record in a diary any changes in medication that occurred during the CFO intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boissy, PhD, Study Director — Université de Sherbrooke; Nathaly Gaudreault, Phd, Study Director — Université de Sherbrooke; Pierre Dagenais, PhD, Study Director — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walha R, Dagenais P, Gaudreault N, Beaudoin-Cote G, Boissy P. The effects of custom-made foot orthoses on foot pain, foot function, gait function, and free-living walking activities in people with psoriatic arthritis (PsA): a pre-experimental trial. Arthritis Res Ther. 2022 May 25;24(1):124. doi: 10.1186/s13075-022-02808-8. PMID 35614481
- [Derived] Walha R, Gaudreault N, Dagenais P, Boissy P. Spatiotemporal parameters and gait variability in people with psoriatic arthritis (PsA): a cross-sectional study. J Foot Ankle Res. 2022 Mar 4;15(1):19. doi: 10.1186/s13047-022-00521-y. PMID 35246222